CLINICAL TRIAL: NCT02368678
Title: Effect Off Full Mouth Disinfection And Scaling Root Planing Per Quadrant In Halitosis in Patients With Advanced Chronic Periodontitis: Randomized Controlled Clinical Trial
Brief Title: "Study of Halitosis in Patients With Advanced Chronic Periodontitis"
Acronym: HACP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Juliana Oliveira da Silveira, Juliana Oliveira da Silveira, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K4gnj9dd
Record Dates: First submitted 2015-02-08; First posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Periodontal Disease; Halitosis; Periodontitis
Keywords: Halitosis; Sulfur compounds; Periodontitis; Periodontal treatment
MeSH Terms: conditions — Periodontal Diseases; Halitosis; Periodontitis | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scaling and Root Planning (SRP) (Active Comparator): Scaling and root planing (SRP) (n=15): the traditional mechanical periodontal therapy consisting of quadrant-wise (30 min. per quadrant) scaling and root planning performed at weekly sessions (one or two weeks of interval between session) and completed within 2 months.
  Interventions: Procedure: Scaling and Root Planning (SRP)
- Full Mouth Scaling (FMS) (Active Comparator): Full mouth scaling (FMS) (n=15): the alternative mechanical periodontal therapy consisting of full-mouth scaling and root planning completed in a single stage within 24 hours; i.e two sessions (60 min. per session) in two consecutive days.
  Interventions: Procedure: Full Mouth Scaling (FMS)

INTERVENTIONS:
Procedure: Scaling and Root Planning (SRP) — Scaling and Root Planing (n=15): quadrant-wise scaling and root planing performed within four weekly session (30 min. per quadrant).
  Oral malodor was measured by organoleptic test and Oral Chroma (Abilit, Osaka Japan) prior to the oral examination, at Baseline and also at 90 days after treatment. Clinical monitoring and tongue coating index were taken at these same times.
  Oral hygiene instructions were given to all participants.
  Arms: Scaling and Root Planning (SRP)
Procedure: Full Mouth Scaling (FMS) — Full Mouth Scaling (n=15): scaling and root planning was performed in a single stage (within 24 hours); two sessions (60 min. per session) in two consecutive days.
  Oral malodor was measured by organoleptic test and Oral Chroma (Abilit, Osaka Japan) prior to the oral examination, at Baseline and also at 90 days after treatment. Clinical monitoring and tongue coating index were taken at these same times.
  Oral hygiene instructions were given to all participants.
  Arms: Full Mouth Scaling (FMS)

SUMMARY:
The objective of this study was to evaluate whether short-term full mouth disinfection protocol could have a greater reduction in the levels of halitosis and volatile sulfur compound or not, when compared to quadrant-wise scaling and root planing

DETAILED DESCRIPTION:
In recent years, several studies have shown that the levels of volatile sulfur compounds are higher in periodontitis patients. However, the relationship between periodontal disease and bad breath is still controversial. Aspects that should be clarified include its relation to periodontitis severity, the influence of risk variables and the subject of the present research, that is treatment choice. To help clinicians and patients when deciding about mechanical periodontal therapy, 30 patients with advanced chronic periodontitis were selected from the periodontics clinic, Dental School, Pontiphical Catholic University of Minas Gerais from April 2013 to May 2014. A complete periodontal clinical examination was performed and the following parameters were recorded: probing depth (PD), clinical attachment level (CAL), bleeding on probing, plaque index, and tongue coating index. Halitosis was assessed by using the organoleptic method and measurements of volatile sulfur compounds (VSC), including hydrogen sulfide (H2S) and methyl mercaptan (CH3SH) by using gas chromatography, at baseline and 90 days after non-surgical periodontal treatment. After periodontal clinical examination, individuals were randomly allocated to full-mouth scaling (FMS) - completed within 24 hours - or to conventional quadrant-wise scaling and root planing (SRP) - completed within 2 months. Halitosis and sulfur gas levels were were statistically compared (Mann-Whitney and Wilcoxon tests, p < 0.05). For inter- and intra-group comparisons regarding categorical variables Chi-square, McNemar, and Fisher exact tests were used. Primary outcome was halitosis changing.

ELIGIBILITY:
Inclusion Criteria:

* age between 35 and 60 years
* presence of at least 20 natural teeth
* diagnosis of chronic periodontitis
* halitosis
* no smokers

Exclusion Criteria:

* smokers or former smokers
* individuals diagnosed with diabetes and / or immunological disorders
* pregnant or lactating / patients with removable partial dentures and / or fixed or removable orthodontic appliance
* systemic use of antibiotics or anti-inflammatory in the last six months
* need for prophylactic use of antibiotics for performing the treatment
* regular use or use in the last six months of any kind of mouthwash
* individuals who underwent periodontal treatment in the 6 months preceding the start of the study

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Halitosis at 3 months | Baseline and 90 days
  Reduction in the number of patients with halitosis and improvement regarding halitosis severity

SECONDARY OUTCOMES:
Change from baseline in clinical attachment level at 3 months | Baseline and 90 days
  Gain of clinical attachment levels (mean values)

CONTACTS AND LOCATIONS:
Overall Officials: Juliana O. da Silveira, Master, Principal Investigator — Federal University of Minas Gerais

REFERENCES:
- [Background] Tanaka M, Yamamoto Y, Kuboniwa M, Nonaka A, Nishida N, Maeda K, Kataoka K, Nagata H, Shizukuishi S. Contribution of periodontal pathogens on tongue dorsa analyzed with real-time PCR to oral malodor. Microbes Infect. 2004 Oct;6(12):1078-83. doi: 10.1016/j.micinf.2004.05.021. PMID 15380777
- [Background] Tangerman A, Winkel EG. Intra- and extra-oral halitosis: finding of a new form of extra-oral blood-borne halitosis caused by dimethyl sulphide. J Clin Periodontol. 2007 Sep;34(9):748-55. doi: 10.1111/j.1600-051X.2007.01116.x. PMID 17716310
- [Background] Tonzetich J, Carpenter PA. Production of volatile sulphur compounds from cysteine, cystine and methionine by human dental plague. Arch Oral Biol. 1971 Jun;16(6):599-607. doi: 10.1016/0003-9969(71)90063-x. No abstract available. PMID 5283484
- [Result] Bollen CM, Beikler T. Halitosis: the multidisciplinary approach. Int J Oral Sci. 2012 Jun;4(2):55-63. doi: 10.1038/ijos.2012.39. PMID 22722640
- [Result] Awano S, Gohara K, Kurihara E, Ansai T, Takehara T. The relationship between the presence of periodontopathogenic bacteria in saliva and halitosis. Int Dent J. 2002 Jun;52 Suppl 3:212-6. doi: 10.1002/j.1875-595x.2002.tb00927.x. PMID 12090455
- [Result] Awano S, Koshimune S, Kurihara E, Gohara K, Sakai A, Soh I, Hamasaki T, Ansai T, Takehara T. The assessment of methyl mercaptan, an important clinical marker for the diagnosis of oral malodor. J Dent. 2004 Sep;32(7):555-9. doi: 10.1016/j.jdent.2004.06.001. PMID 15386861
- [Result] Bosy A, Kulkarni GV, Rosenberg M, McCulloch CA. Relationship of oral malodor to periodontitis: evidence of independence in discrete subpopulations. J Periodontol. 1994 Jan;65(1):37-46. doi: 10.1902/jop.1994.65.1.37. PMID 8133414
- [Result] Bosy A. Oral malodor: philosophical and practical aspects. J Can Dent Assoc. 1997 Mar;63(3):196-201. PMID 9086681
- [Result] Bornstein MM, Kislig K, Hoti BB, Seemann R, Lussi A. Prevalence of halitosis in the population of the city of Bern, Switzerland: a study comparing self-reported and clinical data. Eur J Oral Sci. 2009 Jun;117(3):261-7. doi: 10.1111/j.1600-0722.2009.00630.x. PMID 19583753
- [Result] Coil JM, Yaegaki K, Matsuo T, Miyazaki H. Treatment needs (TN) and practical remedies for halitosis. Int Dent J. 2002 Jun;52 Suppl 3:187-91. doi: 10.1002/j.1875-595x.2002.tb00922.x. PMID 12090450
- [Result] De Boever EH, Loesche WJ. Assessing the contribution of anaerobic microflora of the tongue to oral malodor. J Am Dent Assoc. 1995 Oct;126(10):1384-93. doi: 10.14219/jada.archive.1995.0049. PMID 7594010
- [Result] Faveri M, Hayacibara MF, Pupio GC, Cury JA, Tsuzuki CO, Hayacibara RM. A cross-over study on the effect of various therapeutic approaches to morning breath odour. J Clin Periodontol. 2006 Aug;33(8):555-60. doi: 10.1111/j.1600-051X.2006.00955.x. PMID 16899098
- [Result] Figueiredo LC, Rosetti EP, Marcantonio E Jr, Marcantonio RA, Salvador SL. The relationship of oral malodor in patients with or without periodontal disease. J Periodontol. 2002 Nov;73(11):1338-42. doi: 10.1902/jop.2002.73.11.1338. PMID 12479639
- [Result] Furne J, Majerus G, Lenton P, Springfield J, Levitt DG, Levitt MD. Comparison of volatile sulfur compound concentrations measured with a sulfide detector vs. gas chromatography. J Dent Res. 2002 Feb;81(2):140-3. PMID 11827259
- [Result] Goldberg S, Kozlovsky A, Gordon D, Gelernter I, Sintov A, Rosenberg M. Cadaverine as a putative component of oral malodor. J Dent Res. 1994 Jun;73(6):1168-72. doi: 10.1177/00220345940730060701. PMID 8046106
- [Result] Greenman J, Duffield J, Spencer P, Rosenberg M, Corry D, Saad S, Lenton P, Majerus G, Nachnani S, El-Maaytah M. Study on the organoleptic intensity scale for measuring oral malodor. J Dent Res. 2004 Jan;83(1):81-5. doi: 10.1177/154405910408300116. PMID 14691119
- [Result] Haas AN, Silveira EM, Rosing CK. Effect of tongue cleansing on morning oral malodour in periodontally healthy individuals. Oral Health Prev Dent. 2007;5(2):89-94. PMID 17722433
- [Result] Imai T, Ii H, Yaegaki K, Murata T, Sato T, Kamoda T. Oral malodorous compound inhibits osteoblast proliferation. J Periodontol. 2009 Dec;80(12):2028-34. doi: 10.1902/jop.2009.090208. PMID 19961386
- [Result] Quirynen M, Dadamio J, Van den Velde S, De Smit M, Dekeyser C, Van Tornout M, Vandekerckhove B. Characteristics of 2000 patients who visited a halitosis clinic. J Clin Periodontol. 2009 Nov;36(11):970-5. doi: 10.1111/j.1600-051X.2009.01478.x. Epub 2009 Oct 6. PMID 19811581
- [Result] Lee CH, Kho HS, Chung SC, Lee SW, Kim YK. The relationship between volatile sulfur compounds and major halitosis-inducing factors. J Periodontol. 2003 Jan;74(1):32-7. doi: 10.1902/jop.2003.74.1.32. PMID 12593593
- [Result] Liu XN, Shinada K, Chen XC, Zhang BX, Yaegaki K, Kawaguchi Y. Oral malodor-related parameters in the Chinese general population. J Clin Periodontol. 2006 Jan;33(1):31-6. doi: 10.1111/j.1600-051X.2005.00862.x. PMID 16367853
- [Result] Massler M. Geriatric nutrition: the role of taste and smell in appetite. J Prosthet Dent. 1980 Mar;43(3):247-50. doi: 10.1016/0022-3913(80)90395-9. PMID 6928191
- [Result] Miyazaki H, Sakao S, Katoh Y, Takehara T. Correlation between volatile sulphur compounds and certain oral health measurements in the general population. J Periodontol. 1995 Aug;66(8):679-84. doi: 10.1902/jop.1995.66.8.679. PMID 7473010
- [Result] Morita M, Wang HL. Relationship between sulcular sulfide level and oral malodor in subjects with periodontal disease. J Periodontol. 2001 Jan;72(1):79-84. doi: 10.1902/jop.2001.72.1.79. PMID 11210077
- [Result] Nadanovsky P, Carvalho LB, Ponce de Leon A. Oral malodour and its association with age and sex in a general population in Brazil. Oral Dis. 2007 Jan;13(1):105-9. doi: 10.1111/j.1601-0825.2006.01257.x. PMID 17241439
- [Result] Ng W, Tonzetich J. Effect of hydrogen sulfide and methyl mercaptan on the permeability of oral mucosa. J Dent Res. 1984 Jul;63(7):994-7. doi: 10.1177/00220345840630071701. PMID 6588090
- [Result] Outhouse TL, Fedorowicz Z, Keenan JV, Al-Alawi R. A Cochrane systematic review finds tongue scrapers have short-term efficacy in controlling halitosis. Gen Dent. 2006 Sep-Oct;54(5):352-9; 360, 367-8; quiz 360. PMID 17004573
- [Result] Pedrazzi V, Sato S, de Mattos Mda G, Lara EH, Panzeri H. Tongue-cleaning methods: a comparative clinical trial employing a toothbrush and a tongue scraper. J Periodontol. 2004 Jul;75(7):1009-12. doi: 10.1902/jop.2004.75.7.1009. PMID 15341360
- [Result] Persson S, Edlund MB, Claesson R, Carlsson J. The formation of hydrogen sulfide and methyl mercaptan by oral bacteria. Oral Microbiol Immunol. 1990 Aug;5(4):195-201. doi: 10.1111/j.1399-302x.1990.tb00645.x. PMID 2082242
- [Result] Pham TA, Ueno M, Zaitsu T, Takehara S, Shinada K, Lam PH, Kawaguchi Y. Clinical trial of oral malodor treatment in patients with periodontal diseases. J Periodontal Res. 2011 Dec;46(6):722-9. doi: 10.1111/j.1600-0765.2011.01395.x. Epub 2011 Jul 18. PMID 21762407
- [Result] Quirynen M, Avontroodt P, Soers C, Zhao H, Pauwels M, Coucke W, van Steenberghe D. The efficacy of amine fluoride/stannous fluoride in the suppression of morning breath odour. J Clin Periodontol. 2002 Oct;29(10):944-54. doi: 10.1034/j.1600-051x.2002.291010.x. PMID 12445227
- [Result] Ratcliff PA, Johnson PW. The relationship between oral malodor, gingivitis, and periodontitis. A review. J Periodontol. 1999 May;70(5):485-9. doi: 10.1902/jop.1999.70.5.485. PMID 10368052
- [Result] Roldan S, Herrera D, O'Connor A, Gonzalez I, Sanz M. A combined therapeutic approach to manage oral halitosis: a 3-month prospective case series. J Periodontol. 2005 Jun;76(6):1025-33. doi: 10.1902/jop.2005.76.6.1025. PMID 15948701
- [Result] Rosenberg M, Septon I, Eli I, Bar-Ness R, Gelernter I, Brenner S, Gabbay J. Halitosis measurement by an industrial sulphide monitor. J Periodontol. 1991 Aug;62(8):487-9. doi: 10.1902/jop.1991.62.8.487. PMID 1920015
- [Result] Rosenberg M. Clinical assessment of bad breath: current concepts. J Am Dent Assoc. 1996 Apr;127(4):475-82. doi: 10.14219/jada.archive.1996.0239. PMID 8655868
- [Result] Saito H, Kawaguchi Y. Halitosis prevention campaign: a report of oral health promotion activities in Japan. Int Dent J. 2002 Jun;52 Suppl 3:197-200. doi: 10.1002/j.1875-595x.2002.tb00924.x. PMID 12090452
- [Result] Sanz M, Roldan S, Herrera D. Fundamentals of breath malodour. J Contemp Dent Pract. 2001 Nov 15;2(4):1-17. PMID 12167916
- [Result] Scully C, Porter S, Greenman J. What to do about halitosis. BMJ. 1994 Jan 22;308(6923):217-8. doi: 10.1136/bmj.308.6923.217. No abstract available. PMID 8111254
- [Result] Socransky SS, Haffajee AD. Dental biofilms: difficult therapeutic targets. Periodontol 2000. 2002;28:12-55. doi: 10.1034/j.1600-0757.2002.280102.x. No abstract available. PMID 12013340
- [Result] Soder B, Johansson B, Soder PO. The relation between foetor ex ore, oral hygiene and periodontal disease. Swed Dent J. 2000;24(3):73-82. PMID 11061205
- [Result] Tangerman A, Winkel EG. The portable gas chromatograph OralChroma: a method of choice to detect oral and extra-oral halitosis. J Breath Res. 2008 Mar;2(1):017010. doi: 10.1088/1752-7155/2/1/017010. Epub 2008 Mar 7. PMID 21386154
- [Result] Teughels W, Dekeyser C, Van Essche M, Quirynen M. One-stage, full-mouth disinfection: fiction or reality? Periodontol 2000. 2009;50:39-51. doi: 10.1111/j.1600-0757.2008.00292.x. No abstract available. PMID 19388952
- [Result] Tonzetich J, Ng SK. Reduction of malodor by oral cleansing procedures. Oral Surg Oral Med Oral Pathol. 1976 Aug;42(2):172-81. doi: 10.1016/0030-4220(76)90121-3. PMID 1066599
- [Result] Tonzetich J. Production and origin of oral malodor: a review of mechanisms and methods of analysis. J Periodontol. 1977 Jan;48(1):13-20. doi: 10.1902/jop.1977.48.1.13. PMID 264535
- [Result] Tsai CC, Chou HH, Wu TL, Yang YH, Ho KY, Wu YM, Ho YP. The levels of volatile sulfur compounds in mouth air from patients with chronic periodontitis. J Periodontal Res. 2008 Apr;43(2):186-93. doi: 10.1111/j.1600-0765.2007.01011.x. PMID 18302621
- [Result] Van Tornout M, Dadamio J, Coucke W, Quirynen M. Tongue coating: related factors. J Clin Periodontol. 2013 Feb;40(2):180-5. doi: 10.1111/jcpe.12031. Epub 2012 Dec 20. PMID 23278504
- [Result] Yaegaki K, Sanada K. Volatile sulfur compounds in mouth air from clinically healthy subjects and patients with periodontal disease. J Periodontal Res. 1992 Jul;27(4 Pt 1):233-8. doi: 10.1111/j.1600-0765.1992.tb01673.x. PMID 1640345
- [Result] Kostelc JG, Preti G, Zelson PR, Brauner L, Baehni P. Oral odors in early experimental gingivitis. J Periodontal Res. 1984 May;19(3):303-12. doi: 10.1111/j.1600-0765.1984.tb00821.x. No abstract available. PMID 6235346
- [Result] Krespi YP, Shrime MG, Kacker A. The relationship between oral malodor and volatile sulfur compound-producing bacteria. Otolaryngol Head Neck Surg. 2006 Nov;135(5):671-6. doi: 10.1016/j.otohns.2005.09.036. PMID 17071291
- [Result] van den Broek AM, Feenstra L, de Baat C. A review of the current literature on aetiology and measurement methods of halitosis. J Dent. 2007 Aug;35(8):627-35. doi: 10.1016/j.jdent.2007.04.009. Epub 2007 Jun 6. PMID 17555859
- [Result] Van der Velden U. The Dutch periodontal screening index validation and its application in The Netherlands. J Clin Periodontol. 2009 Dec;36(12):1018-24. doi: 10.1111/j.1600-051X.2009.01495.x. PMID 19929955
- [Result] Yaegaki K, Coil JM. Examination, classification, and treatment of halitosis; clinical perspectives. J Can Dent Assoc. 2000 May;66(5):257-61. PMID 10833869
- [Result] Yaegaki K, Qian W, Murata T, Imai T, Sato T, Tanaka T, Kamoda T. Oral malodorous compound causes apoptosis and genomic DNA damage in human gingival fibroblasts. J Periodontal Res. 2008 Aug;43(4):391-9. doi: 10.1111/j.1600-0765.2007.01052.x. PMID 18942188
- [Result] Winkel EG, Roldan S, Van Winkelhoff AJ, Herrera D, Sanz M. Clinical effects of a new mouthrinse containing chlorhexidine, cetylpyridinium chloride and zinc-lactate on oral halitosis. A dual-center, double-blind placebo-controlled study. J Clin Periodontol. 2003 Apr;30(4):300-6. doi: 10.1034/j.1600-051x.2003.00342.x. PMID 12694427